CLINICAL TRIAL: NCT00034775
Title: Open-Label Trial Exploring A Switching Regimen From Oral Neuroleptics, Other Than Risperidone, To Risperidone Depot Microspheres
Brief Title: A Study to Assess Safety and Tolerabiltiy Associated With a Switch From Oral Antipsychotic Medications to Long-acting Injectable Risperidone in Patients With Schizophrenia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002761
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2011-01

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Schizophrenia; intramuscular injection; antipsychotic agents; risperidone
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The primary purpose of the study is to assess the safety and tolerability of a long-acting injectable formulation of risperidone when switching from an oral antipsychotic in patients with schizophrenia.

DETAILED DESCRIPTION:
For schizophrenia patients taking oral antipsychotic medications, a long-acting injectable formulation of a antipsychotic medication may eliminate the need for daily medication and enhance patient compliance with the treatment regimen. This is an open-label, non-randomized study of a formulation of risperidone (coated microspheres) injected into the muscle at 2 week intervals over 12 weeks in patients with schizophrenia. The study has two phases: during the first 4 weeks, patients continue treatment with their present medication (haloperidol, quetiapine fumarate, or olanzapine); during the second phase of 12 weeks, patients receive the injectable formulation of risperidone, while continuing to receive their present medication for 3 weeks until the risperidone long-acting injectable reaches effective drug levels. For the remainder of the 12-week treatment phase, patients receive only injectable risperidone every 2 weeks. Safety evaluations include the incidence, type, and severity of treatment-emergent adverse events throughout the study; vital signs (pulse, blood pressure), clinical laboratory tests (hematology, biochemistry, urinalysis), electrocardiograms (ECGs), and extrapyramidial symptoms are also monitored at specified intervals. Assessments of effectiveness include the Positive and Negative Syndrome Scale (PANSS) and overall severity of illness measured by the Clinical Global Impression (CGI) scale. The study hypothesis is that long-acting injectible risperidone will be well-tolerated in the treatment of patients with schizophrenia after switching from treatment with an oral antipsychotic. Risperidone injections (25 milligrams[mg]) every 2 weeks for 12 weeks. Investigator may adjust dosage to 37.5mg or 50 mg (maximum) or supplement risperidone injections with risperidone tablets (1mg), according to symptoms and treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia according to Diagnostic and Statistical Manual of Mental Diseases, 4th edition (DSM-IV)
* currently treated with either oral haloperidol, quetiapine fumarate, or olanzapine for 4 months prior to trial entry
* Positive and Negative Syndrome Scale (PANSS) total score of <=80 and score <= 4 on each of the following PANSS items: conceptual disorganization, hallucinatory behavior, suspiciousness, unusual thought content
* body mass index <= 35 at start of study.

Exclusion Criteria:

* Meet DSM-IV criteria for Axis I diagnosis other than schizophrenia or diagnosis of substance dependence (except nicotine or caffeine dependence)
* history of neuroleptic malignant syndrome, a rare psychotropic-drug reaction, which may be characterized by confusion, reduced consciousness, high fever or pronounced muscle stiffness
* history of disease of the central nervous system, such as stroke, Parkinson's disease, Alzheimer's disease, or Huntington's disease
* known hypersensitivity, intolerance, or unresponsiveness to risperidone
* pregnant or nursing females, or those lacking adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2001-08; Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Incidence, type, and severity of treatment-emergent adverse events throughout the treatment period.

SECONDARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale (PANSS) at end of treatment period (Week 12); Extrapyramidal Symptom Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Lindenmayer JP, Eerdekens E, Berry SA, Eerdekens M. Safety and efficacy of long-acting risperidone in schizophrenia: a 12-week, multicenter, open-label study in stable patients switched from typical and atypical oral antipsychotics. J Clin Psychiatry. 2004 Aug;65(8):1084-9. PMID 15323593